CLINICAL TRIAL: NCT00986323
Title: Airsonett Airshower in Allergic Asthma a Double-blind Randomized Multi-centre Trial
Brief Title: Efficacy Study of Temperature Controlled Laminar Airflow (TLA)-Treatment in Perennial Allergic Asthma
Acronym: 4A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Airsonett AB (Industry)
Collaborators: Commitum AB (Industry); Croel AB (Industry)
Responsible Party: Prof. Dr. Chris Anderson, Head of activity, University Hospital, Linkoeping, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Air 3-03; NCT00986388 (obsolete NCT alias); NCT00986622 (obsolete NCT alias); NCT00986726 (obsolete NCT alias); NCT00986934 (obsolete NCT alias)
Record Dates: First submitted 2009-09-27; First posted 2009-09-29 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Asthma
Keywords: Asthma; Temperature controlled Laminar Airflow; TLA; Perennial allergy; Quality of life; Environmental control
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Temeperature controlled Laminar Airflow (Active Comparator): Active treatment with Temperature controlled Laminar Airflow (TLA)
  Interventions: Device: Temperature controlled Laminar Airflow (TLA)
- Placebo TLA (Placebo Comparator): Placebo TLA treatment
  Interventions: Device: Placebo TLA

INTERVENTIONS:
Device: Temperature controlled Laminar Airflow (TLA) — Nocturnal environmental control with Temperature controlled Laminar Airflow (TLA).
  Other Names: Protexo; TLA
  Arms: Temeperature controlled Laminar Airflow
Device: Placebo TLA — Placebo TLA (without filtration and TLA function)
  Arms: Placebo TLA

SUMMARY:
The purpose of this study is to determine whether nocturnal environmental control with Temperature controlled Laminar Airflow (TLA) is effective as add on treatment in patients with perennial allergic asthma.

DETAILED DESCRIPTION:
Exposure to inhaled allergens is a pathogenetic factor in allergic asthma. However, physical, chemical and combined methods aiming to reduce airborne allergen levels have shown little or no effect in reducing asthma symptoms in people who are sensitive to perennial allergens.Aims and objectives: This study aims to investigate treatment with Temperature controled Laminar Airflow (TLA) with a very low particle concentration directed to the breathing zone in subjects with allergic asthma during night sleep. The hypothesis is that the decreased allergen exposure during the night will have an effect on quality of life and bronchial inflammation.

Method: This is a multicentre, double blind, randomized 52 week parallel trial comparing active TLA treatment with Placebo. For ethical reasons the randomization is 2 to 1 for active and placebo treatment, respectively. A 2 weeks run-in period is inserted between inclusion and randomization, during which the patient shall get familiar with the use of the patient asthma diary and to adhere to the requirements of the study participation. First 12 weeks an unchanged maintenance medication will be kept and week 13-52 medication will be modified to obtain asthma control according to international guidelines (GINA). After inclusion, run-in, randomization and baseline measurements active/placebo treatment with AA will be implemented over 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate voluntarily. Willing and able to comply with the study specific procedures. Signed Informed Consent prior to any study procedure.
* Perennial allergic asthma, male and female, age 7 through 70 years, at time of randomization.
* A miniAQLQ/PAQLQ score of ≤ 5.5.
* Sensitive to pet allergen and/or house dust mites as demonstrated by changed to RAST 0.70 or positive skin prick test (wheal reaction similar to histamine control).
* Daily maintenance dose of at least ICS ≥200µg/day of budesonide or ≥100µg/day of fluticasone since at least 6 months
* Features of partly controlled asthma according to GINA

Exclusion Criteria:

* Current smoker (Non-smoker is defined as abstinent since > 1 year). Children: Parents'indoor smoking.
* Participation in another allergen avoidance program
* Participation in drug trial the preceding 3 months
* Multiple chemical sensitivity (e.g. paint, petrol, perfumes) as primary etiology
* Allergen injection or sublingual treatment in the preceding 2 years
* ICS ≥1200µg/day of budesonide or 1000µg/day of fluticasone
* Significant cardiovascular disease
* Participation in the present trial of a family member within the same household

Other protocol-defined exclusion criteria may apply

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2008-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
miniAQLQ (Mini Asthma Quality of Life Questionnaire, Appendix 1) and the corresponding paediatric PAQLQ score. | Week -2, 0, 4, 12, 24, 36 and 52

SECONDARY OUTCOMES:
FENO (Nitric Oxide in Exhaled Air) | Week -2, 0, 4, 12, 24, 36 and 52
Lung function assessed by forced expiratory volume (FEV1), PEF (Expiratory peak flow) and FEF50 (Predicted Forced Expiratory Flow Rate at 50 Percent of Vital Capacity) | Week -2, 0, 4, 12, 24, 36 and 52
Rhinitis symptoms assessed by questionnaire | Week 0 and 52
RAST value and eosinophil count. | Week 0 and 52
Asthma Control Test (ACT). | Week -2, 0, 12, 24, 36 and 52
Resource consumption | Week 0, 4, 12, 24, 36 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Olof Zetterström, MD, PhD., Principal Investigator — University Hospital, Linkoeping
Locations (19):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Bispebjerg Hospital, Copenhagen
- Turku Allergy Centre, Turku, Finland
- Germany (4):
  - Ruhr University of Bochum, Bochum
  - University of München, München
  - University of Rostock, Rostock
  - Marien Hospital Wesel, Wesel
- Norway (2):
  - Ullevaal University Hospital, Oslo
  - St. Olavs Hospital, Trondheim
- Sweden (9):
  - Ängelholm Hospital, Ängelholm
  - Sahlgrenska University Hospital, Sweden, Gothenburg
  - Jonkoping County Hospital, Jönköping
  - County Council of Värmland, Karlstad
  - University Hospital, Linkoeping, Linköping
  - Lund University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - S:t Görans Hospital, Sweden, Stockholm
  - Stockholm South General Hospital, Stockholm
- Imperial College London, London, United Kingdom

REFERENCES:
- [Derived] Boyle RJ, Pedroletti C, Wickman M, Bjermer L, Valovirta E, Dahl R, Von Berg A, Zetterstrom O, Warner JO; 4A Study Group. Nocturnal temperature controlled laminar airflow for treating atopic asthma: a randomised controlled trial. Thorax. 2012 Mar;67(3):215-21. doi: 10.1136/thoraxjnl-2011-200665. Epub 2011 Nov 30. PMID 22131290